CLINICAL TRIAL: NCT00663000
Title: Observational, Cross-sectional, Longitudinal, Multi-center, Diagnostic Study to Evaluate the Influence of Acromegaly on Glucose Tolerance and to Evaluate the Changes of Impaired Glucose Tolerance During Standard Treatment of Acromegaly.
Brief Title: Glucose Tolerance in Acromegaly: The Influence of GH-excess on Glucose Metabolism and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Pfizer (Industry); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Baptist Gallwitz, Prof. Dr. med., University Hospital Tuebingen
Other Study IDs: T-7538; T-7538
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Acromegaly; Diabetes; Insulin Resistance; Impaired Glucose Tolerance
Keywords: acromegaly; diabetes; insulin resistance; impaired glucose tolerance
MeSH Terms: conditions — Acromegaly; Diabetes Mellitus; Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acromegalics: 1. Acromegaly in adult subjects either controlled or uncontrolled (Diagnosis should be based on OGTT where Acromegaly is defined as a lack of suppression of GH nadir to < 0.5 ng/dL, after oral administration of 75 g of glucose, OGTT and IGF-I levels at least 10 % above the normal value ± 2 SD).
  2. Written informed consent

SUMMARY:
Observational, Cross-sectional, longitudinal, multi-center, diagnostic study

Cross-sectional part of the study: To evaluate the influence of acromegaly on glucose tolerance

Longitudinal part of the study: To evaluate the changes of impaired glucose tolerance during standard treatment of acromegaly. Adult patients with established acromegaly

Cross-sectional part of the study: 150 patients

Longitudinal part of the study: 58 patients

DETAILED DESCRIPTION:
TRIAL DESIGN Observational, cross-sectional (patients with normal glucose tolerance). longitudinal (patients with impaired glucose tolerance), multi-center, diagnostic study.

After checking the inclusion and exclusion criteria for the cross-sectional part of the study patients will be included for anamnesis according to Flow Chart Visit -1 (Screening Visit). After checking the glucose tolerance and the insulin resistance by HOMA-IR, the patients will be classified to the group with normal glucose tolerance defined as:

* fasting plasma glucose < 110 mg/dl and/or 2-hour plasma glucose after an OGTT < 140 mg/dl or to the group with impaired glucose tolerance defined as:

  * fasting plasma glucose ≥ 110 mg/dl (IFG) and/or 2-hour plasma glucose after an OGTT ≥ 140 mg/dl (IGT). For the HOMA-IR the cut off is 1.5.

For patients with normal glucose tolerance the study will end after Screening Visit (V -1).

After patient recruitment of the cross-sectional part is completed an interim analysis is planned to verify that all criteria for the longitudinal study part are achieved. The longitudinal part should start not later than one year after the last patient was examined in the cross-sectional part. For patients with impaired glucose tolerance the inclusion and exclusion criteria for the longitudinal part of the study will be checked (Baseline, Visit 0). If a patient might be included into the longitudinal part of the study a 12 months observation with 4 further visits will follow.

Primary Objective and Endpoint

Cross-sectional part of the study:

To evaluate a correlation between IGF-I and glucose tolerance in acromegalic patients. The inclusion should be performed in 2 stratification groups.

Following two groups are defined:

1. 1/3 of patients with a controlled IGF-I (controlled means IGF-I in age and sex-related normal reference range.
2. 2/3 of patients with an uncontrolled IGF-I (uncontrolled means IGF-I not in age and sex related normal reference range.

Longitudinal part of the study:

To evaluate changes of impaired glucose tolerance by different standard treatment options in acromegaly.

For the analysis of the different treatment options patients will be stratified into 5 treatment groups. Decision will be made according to next planned therapeutic intervention at Screening Visit (V -1):

1. Surgery
2. Treatment with somatostatin analoga (with or without combination of dopamine agonists)
3. Treatment with growth hormone receptor antagonist
4. Treatment with somatostatin analoga in combination with growth hormone receptor antagonist
5. Others (e.g. radiation, dopamine agonist monotherapy, no intervention)

ELIGIBILITY:
Inclusion Criteria:

1. Acromegaly in adult subjects (≥ 18 years) either controlled or uncontrolled (Diagnosis should be based on OGTT where Acromegaly is defined as a lack of suppression of GH nadir to < 0.5 ng/dL, after oral administration of 75 g of glucose, OGTT and IGF-I levels at least 10 % above the normal value ± 2 SD).
2. Written informed consent

Exclusion Criteria:

1. Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis, or persistent ALT, AST, alkaline phosphatase 3 x > upper limit of normal, or total bilirubin 2 x > upper limit of normal.
2. Renal failure (GFR ≤ 30 ml/min)
3. Abnormal clinical laboratory values considered by the investigator to be clinically significant and which could affect the interpretation of the study results.
4. History of malignancy of any organ system, treated or untreated, within the past 3 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
5. Suspected or known drug or alcohol abuse.
6. Any condition which in the opinion of the investigator makes the patient unsuitable for inclusion.
7. Participation in any other clinical trial with an investigational new drug.
8. Patients on longterm, continuous (more than 2 weeks/year) systemic therapy with glucocorticosteroids with exception of a substitution of a pituitary lack of ACTH/cortisol (e.g. patients with panhypopituitarism).
9. Instable heart insufficiency for example cardiomyopathy, congestive heart failure (NYHA class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation).
10. Type I diabetes according to the guidelines of the European Diabetes Society or obvious other manifestations of other forms of diabetes (e.g. steroid diabetes).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Acromegaly in adult subjects (≥ 18 years) either controlled or uncontrolled (Diagnosis should be based on OGTT where Acromegaly is defined as a lack of suppression of GH nadir to < 0.5 ng/dL, after oral administration of 75 g of glucose, OGTT and IGF-I levels at least 10 % above the normal value ± 2 SD).
  2. Written informed consent
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate a correlation between IGF-I and glucose tolerance in patients with acromegaly.To evaluate changes of impaired glucose tolerance by different treatment options for acromegaly. | cross-sectional; 1 year longitudinal

SECONDARY OUTCOMES:
Evaluate a correlation between body weight/BMI, age, family history of diabetes,duration of acromegaly and current medical treatment for acromegaly and glucose tolerance / insulin resistance | cross-sectional, 1 year longitudinal

CONTACTS AND LOCATIONS:
Overall Officials: Baptist Gallwitz, MD, Prof., Principal Investigator — Dept. Medicine IV. Tuebingen University
Locations (6):
- Germany (6):
  - Dept. Internal Medicine, Div. Endocrinology, Charité Campus Mitte, University of Berlin, Berlin
  - Endokrinologikum Dresden, Dresden
  - Dept. Internal Medicine, Div. Endocrinology, University of Magdeburg, Magdeburg
  - Dept. Internal Medicine, Endocrinology, Max Planck Institute for Neuroscience and Psychiatry, München
  - Internistische/Endokrinologische Praxis Dr. Droste, Oldenburg
  - Dept. Medicine IV, Tübingen

REFERENCES:
- [Background] Abosch A, Tyrrell JB, Lamborn KR, Hannegan LT, Applebury CB, Wilson CB. Transsphenoidal microsurgery for growth hormone-secreting pituitary adenomas: initial outcome and long-term results. J Clin Endocrinol Metab. 1998 Oct;83(10):3411-8. doi: 10.1210/jcem.83.10.5111. PMID 9768640
- [Background] Abs R, Verhelst J, Maiter D, Van Acker K, Nobels F, Coolens JL, Mahler C, Beckers A. Cabergoline in the treatment of acromegaly: a study in 64 patients. J Clin Endocrinol Metab. 1998 Feb;83(2):374-8. doi: 10.1210/jcem.83.2.4556. PMID 9467544
- [Background] Ahmed S, Elsheikh M, Stratton IM, Page RC, Adams CB, Wass JA. Outcome of transphenoidal surgery for acromegaly and its relationship to surgical experience. Clin Endocrinol (Oxf). 1999 May;50(5):561-7. doi: 10.1046/j.1365-2265.1999.00760.x. PMID 10468920
- [Background] Barkan AL, Halasz I, Dornfeld KJ, Jaffe CA, Friberg RD, Chandler WF, Sandler HM. Pituitary irradiation is ineffective in normalizing plasma insulin-like growth factor I in patients with acromegaly. J Clin Endocrinol Metab. 1997 Oct;82(10):3187-91. doi: 10.1210/jcem.82.10.4249. PMID 9329336
- [Background] Bates AS, Van't Hoff W, Jones JM, Clayton RN. An audit of outcome of treatment in acromegaly. Q J Med. 1993 May;86(5):293-9. PMID 8327647
- [Background] Biermasz NR, van Dulken H, Roelfsema F. Long-term follow-up results of postoperative radiotherapy in 36 patients with acromegaly. J Clin Endocrinol Metab. 2000 Jul;85(7):2476-82. doi: 10.1210/jcem.85.7.6699. PMID 10902796
- [Background] Caron P, Tabarin A, Cogne M, Chanson P, Jaquet P. Variable growth hormone profiles following withdrawal of long-term 30mg slow-release lanreotide treatment in acromegalic patients: clinical implications. Eur J Endocrinol. 2000 Jun;142(6):565-71. doi: 10.1530/eje.0.1420565. PMID 10822218
- [Background] Clemmons DR. Roles of insulin-like growth factor-I and growth hormone in mediating insulin resistance in acromegaly. Pituitary. 2002;5(3):181-3. doi: 10.1023/a:1023321421760. PMID 12812310
- [Background] Colao A, Pivonello R, Auriemma RS, De Martino MC, Bidlingmaier M, Briganti F, Tortora F, Burman P, Kourides IA, Strasburger CJ, Lombardi G. Efficacy of 12-month treatment with the GH receptor antagonist pegvisomant in patients with acromegaly resistant to long-term, high-dose somatostatin analog treatment: effect on IGF-I levels, tumor mass, hypertension and glucose tolerance. Eur J Endocrinol. 2006 Mar;154(3):467-77. doi: 10.1530/eje.1.02112. PMID 16498061
- [Background] Davies PH, Stewart SE, Lancranjan L, Sheppard MC, Stewart PM. Long-term therapy with long-acting octreotide (Sandostatin-LAR) for the management of acromegaly. Clin Endocrinol (Oxf). 1998 Mar;48(3):311-6. doi: 10.1046/j.1365-2265.1998.00389.x. PMID 9578821
- [Background] Eastman RC, Gorden P, Glatstein E, Roth J. Radiation therapy of acromegaly. Endocrinol Metab Clin North Am. 1992 Sep;21(3):693-712. PMID 1521519
- [Background] Elmlinger MW, Kuhnel W, Weber MM, Ranke MB. Reference ranges for two automated chemiluminescent assays for serum insulin-like growth factor I (IGF-I) and IGF-binding protein 3 (IGFBP-3). Clin Chem Lab Med. 2004;42(6):654-64. doi: 10.1515/CCLM.2004.112. PMID 15259383
- [Background] Ezzat S, Forster MJ, Berchtold P, Redelmeier DA, Boerlin V, Harris AG. Acromegaly. Clinical and biochemical features in 500 patients. Medicine (Baltimore). 1994 Sep;73(5):233-40. PMID 7934807
- [Background] Fahlbusch R, Honegger J, Buchfelder M. Evidence supporting surgery as treatment of choice for acromegaly. J Endocrinol. 1997 Oct;155 Suppl 1:S53-5. PMID 9389996
- [Background] Feenstra J, de Herder WW, ten Have SM, van den Beld AW, Feelders RA, Janssen JA, van der Lely AJ. Combined therapy with somatostatin analogues and weekly pegvisomant in active acromegaly. Lancet. 2005 May 7-13;365(9471):1644-6. doi: 10.1016/S0140-6736(05)63011-5. PMID 15885297
- [Background] Feenstra J, van Aken MO, de Herder WW, Feelders RA, van der Lely AJ. Drug-induced hepatitis in an acromegalic patient during combined treatment with pegvisomant and octreotide long-acting repeatable attributed to the use of pegvisomant. Eur J Endocrinol. 2006 Jun;154(6):805-6. doi: 10.1530/eje.1.02160. PMID 16728538
- [Background] Flogstad AK, Halse J, Bakke S, Lancranjan I, Marbach P, Bruns C, Jervell J. Sandostatin LAR in acromegalic patients: long-term treatment. J Clin Endocrinol Metab. 1997 Jan;82(1):23-8. doi: 10.1210/jcem.82.1.3572. PMID 8989226
- [Background] Giustina A, Barkan A, Casanueva FF, Cavagnini F, Frohman L, Ho K, Veldhuis J, Wass J, Von Werder K, Melmed S. Criteria for cure of acromegaly: a consensus statement. J Clin Endocrinol Metab. 2000 Feb;85(2):526-9. doi: 10.1210/jcem.85.2.6363. PMID 10690849
- [Background] Hansen I, Tsalikian E, Beaufrere B, Gerich J, Haymond M, Rizza R. Insulin resistance in acromegaly: defects in both hepatic and extrahepatic insulin action. Am J Physiol. 1986 Mar;250(3 Pt 1):E269-73. doi: 10.1152/ajpendo.1986.250.3.E269. PMID 3513613
- [Background] Hunter SJ, Shaw JA, Lee KO, Wood PJ, Atkinson AB, Bevan JS. Comparison of monthly intramuscular injections of Sandostatin LAR with multiple subcutaneous injections of octreotide in the treatment of acromegaly; effects on growth hormone and other markers of growth hormone secretion. Clin Endocrinol (Oxf). 1999 Feb;50(2):245-51. doi: 10.1046/j.1365-2265.1999.00668.x. PMID 10396369
- [Background] Jaffe CA, Barkan AL. Treatment of acromegaly with dopamine agonists. Endocrinol Metab Clin North Am. 1992 Sep;21(3):713-35. PMID 1355728
- [Background] Jorgensen JO, Feldt-Rasmussen U, Frystyk J, Chen JW, Kristensen LO, Hagen C, Orskov H. Cotreatment of acromegaly with a somatostatin analog and a growth hormone receptor antagonist. J Clin Endocrinol Metab. 2005 Oct;90(10):5627-31. doi: 10.1210/jc.2005-0531. Epub 2005 Jul 26. PMID 16046586
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Melmed S. Acromegaly. N Engl J Med. 1990 Apr 5;322(14):966-77. doi: 10.1056/NEJM199004053221405. No abstract available. PMID 2179724
- [Background] Moller N, Schmitz O, Joorgensen JO, Astrup J, Bak JF, Christensen SE, Alberti KG, Weeke J. Basal- and insulin-stimulated substrate metabolism in patients with active acromegaly before and after adenomectomy. J Clin Endocrinol Metab. 1992 May;74(5):1012-9. doi: 10.1210/jcem.74.5.1569148.
- [Background] Orme SM, McNally RJ, Cartwright RA, Belchetz PE. Mortality and cancer incidence in acromegaly: a retrospective cohort study. United Kingdom Acromegaly Study Group. J Clin Endocrinol Metab. 1998 Aug;83(8):2730-4. doi: 10.1210/jcem.83.8.5007. PMID 9709939
- [Background] Osman IA, James RA, Chatterjee S, Mathias D, Kendall-Taylor P. Factors determining the long-term outcome of surgery for acromegaly. QJM. 1994 Oct;87(10):617-23. PMID 7987657
- [Background] Rajasoorya C, Holdaway IM, Wrightson P, Scott DJ, Ibbertson HK. Determinants of clinical outcome and survival in acromegaly. Clin Endocrinol (Oxf). 1994 Jul;41(1):95-102. doi: 10.1111/j.1365-2265.1994.tb03789.x. PMID 8050136
- [Background] Rose DR, Clemmons DR. Growth hormone receptor antagonist improves insulin resistance in acromegaly. Growth Horm IGF Res. 2002 Dec;12(6):418-24. doi: 10.1016/s1096-6374(02)00083-7. PMID 12423627
- [Background] Sacca L, Cittadini A, Fazio S. Growth hormone and the heart. Endocr Rev. 1994 Oct;15(5):555-73. doi: 10.1210/edrv-15-5-555. PMID 7843068
- [Background] Schreiber I, Buchfelder M, Droste M, Forssmann K, Mann K, Saller B, Strasburger CJ; German Pegvisomant Investigators. Treatment of acromegaly with the GH receptor antagonist pegvisomant in clinical practice: safety and efficacy evaluation from the German Pegvisomant Observational Study. Eur J Endocrinol. 2007 Jan;156(1):75-82. doi: 10.1530/eje.1.02312. PMID 17218728
- [Background] Stumvoll M, Van Haeften T, Fritsche A, Gerich J. Oral glucose tolerance test indexes for insulin sensitivity and secretion based on various availabilities of sampling times. Diabetes Care. 2001 Apr;24(4):796-7. doi: 10.2337/diacare.24.4.796. No abstract available. PMID 11315860
- [Background] Sze L, Schmid C, Bloch KE, Bernays R, Brandle M. Effect of transsphenoidal surgery on sleep apnoea in acromegaly. Eur J Endocrinol. 2007 Mar;156(3):321-9. doi: 10.1530/eje.1.02340. PMID 17322492
- [Background] Swearingen B, Barker FG 2nd, Katznelson L, Biller BM, Grinspoon S, Klibanski A, Moayeri N, Black PM, Zervas NT. Long-term mortality after transsphenoidal surgery and adjunctive therapy for acromegaly. J Clin Endocrinol Metab. 1998 Oct;83(10):3419-26. doi: 10.1210/jcem.83.10.5222. PMID 9768641
- [Background] Tindall GT, Oyesiku NM, Watts NB, Clark RV, Christy JH, Adams DA. Transsphenoidal adenomectomy for growth hormone-secreting pituitary adenomas in acromegaly: outcome analysis and determinants of failure. J Neurosurg. 1993 Feb;78(2):205-15. doi: 10.3171/jns.1993.78.2.0205. PMID 8421204
- [Background] van der Lely AJ, de Herder WW, Lamberts SW. A risk-benefit assessment of octreotide in the treatment of acromegaly. Drug Saf. 1997 Nov;17(5):317-24. doi: 10.2165/00002018-199717050-00004. PMID 9391775
- [Background] van der Lely AJ, Muller A, Janssen JA, Davis RJ, Zib KA, Scarlett JA, Lamberts SW. Control of tumor size and disease activity during cotreatment with octreotide and the growth hormone receptor antagonist pegvisomant in an acromegalic patient. J Clin Endocrinol Metab. 2001 Feb;86(2):478-81. doi: 10.1210/jcem.86.2.7206. PMID 11157994
- [Background] Veysey MJ, Thomas LA, Mallet AI, Jenkins PJ, Besser GM, Wass JA, Murphy GM, Dowling RH. Prolonged large bowel transit increases serum deoxycholic acid: a risk factor for octreotide induced gallstones. Gut. 1999 May;44(5):675-81. doi: 10.1136/gut.44.5.675. PMID 10205204
- [Background] Wasada T, Aoki K, Sato A, Katsumori K, Muto K, Tomonaga O, Yokoyama H, Iwasaki N, Babazono T, Takahashi C, Iwamoto Y, Omori Y, Hizuka N. Assessment of insulin resistance in acromegaly associated with diabetes mellitus before and after transsphenoidal adenomectomy. Endocr J. 1997 Aug;44(4):617-20. doi: 10.1507/endocrj.44.617. PMID 9447299